CLINICAL TRIAL: NCT00048204
Title: An 8-Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Fixed-Dose Study Comparing the Efficacy and Safety of GW597599B or Paroxetine to Placebo in Moderately to Severely Depressed Patients With Major Depressive Disorder
Brief Title: A Study Of A New Medicine (GW597599B) For The Treatment Of Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKD20006
Record Dates: First submitted 2002-10-28; First posted 2002-10-30 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Psychiatry; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW597599B
Drug: paroxetine
  Other Names: GW597599B

SUMMARY:
A Placebo Controlled Study Evaluating Efficacy And Safety of Medication In Patients With Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Patients meet the diagnosis of Major Depressive Disorder (MDD).

Exclusion Criteria:

* Patients with a primary diagnosis other than MDD.
* Patients with a history of schizophrenia, schizoaffective disorders, seizure disorders or bipolar affective disorder.
* Patients receiving formal psychotherapy or cognitive/behavioral therapy concurrently or in the 12 weeks prior to screening visit.
* Patient is actively suicidal.
* Patients who have a history of migraine headaches.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2002-11-04 (Actual); Primary Completion 2003-09-30 (Actual); Study Completion 2003-09-30

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 8 Weeks

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale Clinical Global Impression-Global Improvement Clinical Global Impression-Severity of Illness Hospital Anxiety and Depression Scale | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKD20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register